CLINICAL TRIAL: NCT00279786
Title: B2-Adrenergic Receptor Polymorphisms: Implications For The Treatment Of Status Asthmaticus In Children
Brief Title: B2-Adrenergic Receptor Polymorphisms
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-001
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2009-07

CONDITIONS: Status Asthmaticus
Keywords: pediatric
MeSH Terms: conditions — Status Asthmaticus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood draw — blood drawn
  Other Names: genotyping of ß2-AR at position 16 and 27.

SUMMARY:
Beta(2)-adrenergic receptor (BAR) agonists are the most important group of drugs used in the treatment of asthma. In children unresponsive to inhaled BAR agonist therapy, higher dose systemic BAR agonist therapy is frequently the next step in treatment. Despite the widespread use of intravenous BAR agonist therapy for pediatric status asthmaticus, there is controversy regarding the efficacy of this therapy. A number of studies have established that genetic variations of the BAR have important effects in modulating responses to BAR agonist therapy for asthma. In particular, changes in amino acid position 16 of the BAR gene are thought to be the most functionally important. Patients encoded for two glycine amino acids, rather than arginine, at this position appear to have more severe asthma and to respond differently to acute BAR agonist therapy.

Our hypothesis is that genotypic differences may contribute to poor response to acute BAR agonist treatment. We propose to conduct a prospective observational study to determine the influence of a patient's BAR genotype on the response to acute BAR agonist therapy.

Our specific hypothesis is that children with genetic polymorphisms of the gene encoding the BAR will have a decreased response to acute high-dose continuous BAR therapy (both inhaled and intravenous) compared to other children.

Our primary outcome is ICU length of stay. Secondary outcomes are

1. to assess the rate of improvement in clinical asthma score based on genotype, and
2. to attempt to correlate asthma phenotype with genotype by comparing demographic data and hospital course.

DETAILED DESCRIPTION:
This study has both a prospective and a retrospective arm. In the retrospective arm, patients with a history of admission to the ICU with a severe asthma exacerbation are contacted by phone and mail and DNA samples are obtained via saliva. In the prospective arm, patients admitted to the ICU are contacted prospectively and DNA is obtained either via saliva or blood.

ELIGIBILITY:
Inclusion Criteria:

* (1) Admission to the CCMC PICU with a primary admission diagnosis of status asthmaticus. (2) Age between 2 years and 18 years.

Exclusion Criteria:

* Pre-existing chronic disease (other than asthma)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to the ICU with severe asthma exacerbations
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2005-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carroll, MD, Principal Investigator — CT Children's Medical Center
Locations (1):
- CT Children's Medical Center, Hartford, Connecticut, United States